CLINICAL TRIAL: NCT01227369
Title: Quality of Life(QoL) in Korean Postmenopausal Osteoporosis Patients With Bisphosphonate Treatment
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111720
Record Dates: First submitted 2010-06-03; First posted 2010-10-25 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Bisphosphonates; OPSAT-Q
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bisphosphonates: Korean postmenopausal osteoporosis patients with bisphosphonate treatment
  Interventions: Other: OPSAT-Q

INTERVENTIONS:
Other: OPSAT-Q — A linguistically validated Korean version of OPSAT-Q

SUMMARY:
Quality of Life (QoL) in Korean postmenopausal osteoporosis patients with bisphosphonate treatment

DETAILED DESCRIPTION:
Cross-sectional quality of life survey using self-administered OPSAT-QTM questionnaire in Korean postmenopausal osteoporosis patients with bisphosphonate treatment

ELIGIBILITY:
Inclusion Criteria:

* Who have been diagnosed with postmenopausal osteoporosis by physician Who have received any oral bisphosphonates (weekly or monthly) at least for 2 months to provide answer of OPSAT-QTM questionnaire Who provide informed consent for study participation

Exclusion Criteria:

* Do not understand the contents of the questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to 2006 national health insurance data, a total of osteoporosis women (ICD-10 code: M81) are about 244,190 in Korea According to recent market research data, 95% of osteoporosis women use bisphosphonate in Korea.
  With considering 95% market share of bisphosphonate in osteoporosis market, there are 231,714 Korean osteoporosis women. Applying for 2% extracting fraction in this study, total size of study population are 4,634.
Sampling Method: Probability Sample
Enrollment: 4376 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Mean of composite satisfaction score (CSS) of OPSAT-QTM | 0day

SECONDARY OUTCOMES:
Mean of subscale satisfaction scores of OPSAT-QTM | oday

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea